CLINICAL TRIAL: NCT02799381
Title: An Open-label, Randomized 12 Week Study Comparing Efficacy of Levodopa-Carbidopa Intestinal Gel/Carbidopa-Levodopa Enteral Suspension and Optimized Medical Treatment on Dyskinesia in Subjects With Advanced Parkinson's Disease DYSCOVER (DYSkinesia COmparative Interventional Trial on Duodopa VERsus Oral Medication)
Brief Title: A Study Comparing Efficacy of Levodopa-Carbidopa Intestinal Gel/Carbidopa-Levodopa Enteral Suspension and Optimized Medical Treatment on Dyskinesia in Subjects With Advanced Parkinson's Disease (DYSCOVER)
Acronym: DYSCOVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-535; 2016-001403-23 (EudraCT Number)
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Parkinson's Disease (PD)
Keywords: Carbidopa; Levodopa; Efficacy; Levodopa-carbidopa intestinal gel; Advanced Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimized Medical Treatment (OMT) (Active Comparator): Participants randomized to OMT continued their current anti Parkinson's disease (anti-PD) medication regimen for the duration of the study. All anti-PD medications and medications to treat dyskinesia must have remained stable for the duration of the study unless adjustments were medically indicated. The Investigator provided the prescription for continued OMT.
  Interventions: Drug: Optimized antiparkinsonian treatment
- Levodopa-Carbidopa Intestinal Gel (LCIG) (Experimental): The total daily dose of infusion LCIG was composed of three components: (i) the morning dose, (ii) continuous maintenance infusion dose and (iii) extra doses. A temporary nasojejunal (NJ) tube may have been used initially with the infusion pump to determine a participant's response to this method of treatment and to optimize the dose of LCIG before treatment with a permanent percutaneous endoscopic gastrostomy - with jejunal extension (PEG-J) tube was started. Following optional NJ and/or PEG-J placement and, at the investigator's discretion, the participant may have begun initiation and titration of LCIG infusion on Day 1 once tube placement was confirmed. The dose of LCIG was adjusted to obtain the optimal clinical response. The rate of LCIG infusion is typically within the range of 1 to 10 mL/hour (20 to 200 mg of levodopa/hour) in most instances and runs over a period of 16 consecutive hours each day.
  Interventions: Drug: Levodopa-Carbidopa Intestinal Gel (LCIG); Device: CADD-Legacy ambulatory infusion pump; Device: Percutaneous endoscopic gastrostomy tube; Device: Jejunal extension tube

INTERVENTIONS:
Drug: Optimized antiparkinsonian treatment — Dose levels of prescribed antiparkinsonian medications were individually optimized to their maximum therapeutic effect.
  Arms: Optimized Medical Treatment (OMT)
Drug: Levodopa-Carbidopa Intestinal Gel (LCIG) — Dose levels were individually optimized.
  Other Names: ABT-SLV187; DUOPA (carbidopa and levodopa Enteral Suspension); DUODOPA
  Arms: Levodopa-Carbidopa Intestinal Gel (LCIG)
Device: CADD-Legacy ambulatory infusion pump — (manufactured by Smiths Medical)
  Arms: Levodopa-Carbidopa Intestinal Gel (LCIG)
Device: Percutaneous endoscopic gastrostomy tube — (PEG tube)
  Arms: Levodopa-Carbidopa Intestinal Gel (LCIG)
Device: Jejunal extension tube — (J-tube)
  Arms: Levodopa-Carbidopa Intestinal Gel (LCIG)

SUMMARY:
The primary objective of this study was to examine the effect of levodopa-carbidopa intestinal gel (LCIG) compared with optimized medical treatment (OMT) on dyskinesia in participants with advanced Parkinson's disease (PD).

DETAILED DESCRIPTION:
This was a Phase 3b, open-label, randomized, multicenter, 12-week study. The study consisted of 3 sequential periods: Screening, Treatment, and Follow-Up. The OMT group had the same schedule of visits/procedures throughout the study as the LCIG treatment group, except for visits related to nasojejunal (NJ)/percutaneous endoscopic gastrostomy (PEG) procedures, titration of LCIG, and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of idiopathic Parkinson's disease (PD) according to the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria
* Participants with advanced levodopa-responsive PD and persistent motor fluctuations who have not been controlled with optimized medical treatment (OMT: the maximum therapeutic effect obtained with pharmacological antiparkinsonian therapies when no further improvement is expected with regard to any additional manipulations of levodopa and/or other antiparkinsonian medication based on the Investigator's clinical judgment)
* Unified Dyskinesia Rating Scale (UDysRs) Total score ≥ 30 at Visit 3

Exclusion Criteria:

* Participant(s) treated with levodopa-carbidopa intestinal gel (LCIG) previously
* Participant's PD diagnosis is unclear or there is a suspicion that the subject has a parkinsonian syndrome such as secondary parkinsonism (e.g. caused by drugs, toxins, infectious agents, vascular disease, trauma, brain neoplasm), parkinson-plus syndrome (e.g. Multiple System Atrophy, Progressive supranuclear Palsy, Diffuse Lewy Body disease) or other neurodegenerative disease that might mimic the symptoms of PD
* Participant(s) has undergone neurosurgery for the treatment of Parkinson's disease.
* Participant(s) has contraindications to levodopa (e.g. narrow angle glaucoma, malignant melanoma)
* Participant(s) experiencing clinically significant sleep attacks or clinically significant impulsive behavior (e.g. pathological gambling, hypersexuality) at any point during the three months prior to the Screening evaluation as judged by the Principal Investigator

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (28):
- United States (2):
  - Parkinson's Disease Treatment Center of Southwest Florida /ID# 150095, Port Charlotte, Florida
  - Central Texas Neurology Consul /ID# 150088, Round Rock, Texas
- Finland (2):
  - Helsinki Univ Central Hospital /ID# 151214, Helsinki
  - Oulun yliopistollinen sairaala /ID# 150947, Oulu
- Greece (3):
  - Mediterraneo Hospital /ID# 150955, Glyfada
  - University General Hospital of Heraklion "PA.G.N.I" /ID# 150956, Heraklion
  - University Hospital of Ioannin /ID# 150954, Ioannina
- Hungary (3):
  - Pecsi Tudomanyegyetem Klinikai Kozpont I. sz. Belgyogyaszati Klinika /ID# 170116, Pécs, Pecs
  - Semmelweis Egyetem /ID# 170117, Budapest
  - Szegedi Tudomanyegyetem /ID# 170115, Szeged
- Italy (5):
  - Policlinico Universitario Campus Bio-Medico /ID# 150846, Rome, Lazio
  - A.O. Univ. Ospedali Riuniti /ID# 150853, Ancona, The Marches
  - Azienda USL Toscana Centro /ID# 150770, Florence
  - Seconda Universita' di Napoli /ID# 150851, Naples
  - Policlinico Tor Vergata /ID# 151167, Rome
- Slovakia (4):
  - Univerzitna nemocnica L. Pasteura /ID# 150146, Košice - Západ, Košice Region
  - Univerzitna Nemocnica Bratislava /ID# 150144, Bratislava
  - Univerzitna Nemocnica Bratislava /ID# 150171, Bratislava
  - Univerzitna nemocnica Martin /ID# 150145, Martin, Žilina Region
- Spain (9):
  - Hospital Regional Universitari /ID# 171485, Málaga, Malaga
  - Hospital Universitario Cruces /ID# 203807, Barakaldo
  - Hospital General Univ de Elche /ID# 150154, Elche
  - Hospital Univ de la Princesa /ID# 150157, Madrid
  - Hospital General Universitario Gregorio Maranon /ID# 150155, Madrid
  - Hospital Univ Ramon y Cajal /ID# 150152, Madrid
  - Hospital Universitario Infanta /ID# 159696, Madrid
  - Hospital Universitario Virgen Macarena /ID# 158861, Seville
  - Hospital Virgen de la Salud /ID# 166297, Toledo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Freire-Alvarez E, Vanni P, Kurca E, Lopez-Manzanares L, Kovacs N, Spanaki C, Gao T, Bergmann L, Sanchez-Solino O. Dyskinesia and Pain in Advanced Parkinson's Disease: Post Hoc Analysis from the Phase 3b, Open-Label, Randomized DYSCOVER Study. Neurol Ther. 2024 Apr;13(2):437-447. doi: 10.1007/s40120-024-00583-z. Epub 2024 Feb 12. PMID 38345741
- [Derived] Freire-Alvarez E, Kurca E, Lopez Manzanares L, Pekkonen E, Spanaki C, Vanni P, Liu Y, Sanchez-Solino O, Barbato LM. Levodopa-Carbidopa Intestinal Gel Reduces Dyskinesia in Parkinson's Disease in a Randomized Trial. Mov Disord. 2021 Nov;36(11):2615-2623. doi: 10.1002/mds.28703. Epub 2021 Jul 8. PMID 34236101
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety Data Set: all participants randomized to OMT and all participants randomized to LCIG treatment who had a study tube (NJ or PEG-J) placement procedure. Two participants randomized to the LCIG arm did not have device placement for LCIG infusion and were not included in the safety data set.
Period: Overall Study
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Started | 33 | 28
Completed | 29 | 25
Not Completed | 4 | 3
Not completed — Withdrew consent | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Participant did not take any study drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Data Set: all participants randomized to OMT and all participants randomized to LCIG treatment who had a study tube (NJ or PEG-J) placement procedure. Two participants randomized to the LCIG arm did not have device placement for LCIG infusion and were not included in the safety data set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG) | Total
Number analyzed (Participants) | 33 | 28 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (7.20) | 69.3 (6.99) | 69.0 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 17 | 12 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 28 | 61
  Black or African American | 0 | 0 | 0
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Missing | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (4.42) | 24.5 (4.24) | 24.9 (4.32)
Parkinson's disease duration (years) [Count of Participants; unit: Participants]
  < 10 years | 14 | 7 | 21
  ≥ 10 years | 19 | 20 | 39
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 12 in Unified Dyskinesia Rating Scale (UDysRS) Total Score
Description: The Unified Dyskinesia Rating Scale (UDysRS) is a tool used to assess dyskinesia in Parkinson's disease (PD) and contains both self-evaluation questions and items that are assessed directly by the physician to objectively rate the abnormal movements associated with PD. Part 1 contains 11 questions about the ON time dyskinesia and the impact of ON-dyskinesia on experiences of daily living. Part 2 contains 4 questions about OFF-dystonia rating. Part 3 contains 7 questions about objective evaluation of dyskinesia impairment and Part 4 contains 4 questions regarding dyskinesia disability. Each question is scored with respect to severity, which is rated on a scale where 0 = normal, 1 = slight, 2 = mild, 3= moderate and 4 = severe. The UDysRS total score is obtained by summing the item scores, ranging from 0 to 104. Higher scores are associated with more disability. Negative changes from baseline indicate improvement.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) population: all participants with available data who were randomized to the OMT and all participants who were randomized to LCIG treatment and received at least 1 dose of study drug following PEG-J placement
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 26 | 24
units on a scale | -2.33 (2.56) | -17.37 (2.79)
Statistical Analysis 1: Comparison: Optimized Medical Treatment (OMT) vs Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority — The likelihood-based mixed-effects model repeated measures (MMRM) analysis of the change from baseline to Week 12 used all observed data. The model included fixed, categorical effects for treatment, country, visit, and treatment-by-visit interaction, with continuous fixed covariates for baseline score and the baseline score-by-visit interaction; p < 0.0001, Mixed-effects model repeated measures — Two-sided p-value; LS Mean Difference = -15.05, 95% CI 2-sided [-21.47 to -8.63] — Levodopa-Carbidopa Intestinal Gel (LCIG) - Optimized Medical Treatment (OMT) at Week 12

2. Secondary Outcome: Mean Change From Baseline to Week 12 in ON Time Without Troublesome Dyskinesia
Description: The Parkinson's Disease (PD) Symptom Diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected study visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e., 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. ON time is when PD symptoms are well controlled by the drug, and OFF time is when PD symptoms are not adequately controlled by the drug. Positive change from baseline for ON time without troublesome dyskinesia indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 28 | 25
hours | -0.12 (0.63) | 3.15 (0.69)
Statistical Analysis 1: Comparison: Optimized Medical Treatment (OMT) vs Levodopa-Carbidopa Intestinal Gel (LCIG); If the primary efficacy variable was statistically significant, each of the secondary variables were to be tested using a fixed sequence as a gatekeeping procedure and at α level of 0.050. Testing was to cease at the point that a secondary variable failed to demonstrate statistical significance; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed-effects model repeated measures — Two-sided p-value; LS Mean Difference = 3.27, 95% CI 2-sided [1.71 to 4.83] — Levodopa-Carbidopa Intestinal Gel (LCIG) - Optimized Medical Treatment (OMT) at Week 12

3. Secondary Outcome: Mean Change From Baseline to Week 12 in Parkinson's Disease Questionnaire-8 (PDQ-8) Summary Index
Description: The Parkinson's Disease Questionnaire-8 (PDQ-8) is a disease-specific instrument designed to measure aspects of health that are relevant to participants with PD, and which may not be included in general health status questionnaires. The PDQ-8 is a self-administered questionnaire. Each item is scored on the following 5-point scale: 0 = Never, 1 = Occasionally, 2 = Sometimes, 3 = Often, 4 = Always (or cannot do at all, if applicable). Higher scores are consistently associated with the more severe symptoms of the disease such as tremors and stiffness. The results are presented as a summary index. The PDQ-8 summary index ranges from 0 to 100, where lower scores indicate a better perceived health status. Negative changes from baseline indicate improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29 | 25
units on a scale | -4.95 (3.11) | -21.62 (3.47)
Statistical Analysis 1: Comparison: Optimized Medical Treatment (OMT) vs Levodopa-Carbidopa Intestinal Gel (LCIG); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed-effects model repeated measures — Two-sided p-value; LS Mean Difference = -16.66, 95% CI 2-sided [-24.48 to -8.85] — Levodopa-Carbidopa Intestinal Gel (LCIG) - Optimized Medical Treatment (OMT) at Week 12

4. Secondary Outcome: Mean Clinical Global Impression of Change (CGI-C) Score at Week 12
Description: The Clinical Global Impression of Change (CGI-C) score is a clinician's rating scale for assessing Global Improvement of Change. The CGI-C rates improvement by 7 categories: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), very much worse (7). The CGI-C score ranges from 1 to 7, with lower scores indicating improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 32 | 27
units on a scale | 4.58 (0.25) | 2.48 (0.28)
Statistical Analysis 1: Comparison: Optimized Medical Treatment (OMT) vs Levodopa-Carbidopa Intestinal Gel (LCIG); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed-effects model repeated measures — Two-sided p-value; LS Mean Difference = -2.11, 95% CI 2-sided [-2.78 to -1.44] — Levodopa-Carbidopa Intestinal Gel (LCIG) - Optimized Medical Treatment (OMT) at Week 12

5. Secondary Outcome: Mean Change From Baseline to Week 12 in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score (Activities of Daily Living)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to the 13 questions related to Activities of Daily Living, and ranges from 0-52. Higher scores are associated with more disability. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29 | 24
units on a scale | 0.21 (1.16) | -5.33 (1.28)
Statistical Analysis 1: Comparison: Optimized Medical Treatment (OMT) vs Levodopa-Carbidopa Intestinal Gel (LCIG); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0006, Mixed-effects model repeated measures — Two-sided p-value; LS Mean Difference = -5.54, 95% CI 2-sided [-8.59 to -2.49] — Levodopa-Carbidopa Intestinal Gel (LCIG) - Optimized Medical Treatment (OMT) at Week 12

6. Secondary Outcome: Mean Change From Baseline to Week 12 in OFF Time
Description: The Parkinson's Disease (PD) Symptom Diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected study visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e., 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. ON time is when PD symptoms are well controlled by the drug, and OFF time is when PD symptoms are not adequately controlled by the drug. Negative change from baseline for OFF time indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 28 | 25
hours | 0.18 (0.49) | -2.17 (0.53)
Statistical Analysis 1: Comparison: Optimized Medical Treatment (OMT) vs Levodopa-Carbidopa Intestinal Gel (LCIG); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0002, Mixed-effects model repeated measures — Two-sided p-value; LS Mean Difference = -2.35, 95% CI 2-sided [-3.51 to -1.19] — Levodopa-Carbidopa Intestinal Gel (LCIG) - Optimized Medical Treatment (OMT) at Week 12

7. Secondary Outcome: Mean Change From Baseline to Week 12 in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score (Motor Examination)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part III score is the sum of the 27 answers related to Motor Examination, and ranges from 0-108. Higher scores are associated with more disability. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Optimized Medical Treatment (OMT) | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29 | 25
units on a scale | -0.87 (1.89) | -4.93 (2.08)
Statistical Analysis 1: Comparison: Optimized Medical Treatment (OMT) vs Levodopa-Carbidopa Intestinal Gel (LCIG); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0762, Mixed-effects model repeated measures — Two-sided p-value; LS Mean Difference = -4.05, 95% CI 2-sided [-8.55 to 0.44] — Levodopa-Carbidopa Intestinal Gel (LCIG) - Optimized Medical Treatment (OMT) at Week 12

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) collection: OMT (starting after the day of randomization until 30 days after the last visit, up to 18 weeks); LCIG group with study tube removal after the last study drug infusion (from the time of tube placement up to 30 days following tube removal, up to 16 weeks); other LCIG participants (starting with tube placement and up to 30 days following the last study visit, up to 16 weeks)
Description: TEAEs and SAEs are defined as any adverse event (AE) with an onset date starting after the day of randomization (OMT group) or from the time of tube placement (LCIG group) until 30 days after the last visit (OMT group), or up to 30 days following tube removal (LCIG group) or the last study visit (LCIG group) and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG) | Optimized Medical Treatment (OMT)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/33
Other Adverse Events (participants affected / at risk) | 15/28 | 4/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (LCIG) (N=28) | Optimized Medical Treatment (OMT) (N=33)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (LCIG) (N=28) | Optimized Medical Treatment (OMT) (N=33)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
DRUG WITHDRAWAL SYNDROME (General disorders) | 2 (2) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 6 (6) | 2 (3)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 2 (2)
ANXIETY (Psychiatric disorders) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT02799381/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02799381/SAP_001.pdf